CLINICAL TRIAL: NCT00521937
Title: A Prospective, Randomised, Multi-centre, Blind-observer, Controlled, Parallel-group Study Comparing the Efficacy and Safety of DERMAGEN® Versus Conventional Treatment in the Treatment of Diabetic Neuropathic Foot Ulcer
Brief Title: Efficacy and Safety Study of DERMAGEN® vs Conventional Treatment to Treat Diabetic Neuropathic Foot Ulcer
Acronym: DERMAGEN®
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Laboratoires Genévrier (Industry)
Responsible Party: Fabien AUDIBERT, Laboratoires Genevrier
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06FB/DE02
Record Dates: First submitted 2007-08-27; First posted 2007-08-28 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: Diabetes; Foot Ulcer
MeSH Terms: conditions — Diabetes Mellitus; Foot Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Dermagen®
  Interventions: Other: Dermagen®
- B (Active Comparator): Conventional treatment
  Interventions: Other: Dermagen®

INTERVENTIONS:
Other: Dermagen® — Weekly topical applications

SUMMARY:
It is estimated that 300 million people worldwide will have diabetes by the year 2025. About 12 percent of those with diabetes will have had a foot ulcer, which is a major source of morbidity, concern, and cost.

The foot ulcers are the leading cause of hospitalization among people with diabetes and often lead to amputation. The costs of treatment and the high morbidity and mortality associated with diabetic foot problems necessitate the need for a systemic approach to a foot ulcer management.

Current local treatments of this type of ulcer are: dressings (hydrocolloids, alginate…), and growth factors. However modern dressings may not avoid infection and the results of the clinical studies are not significant in terms of complete healing rate or in terms of time to healing. Concerning growth factors, the only one whose therapeutic application made proof is the rhPDGF (Regranex®) with an increase in the number of ulcers completely healed at the twentieth week compared to placebo (50% and 35%, respectively).

The advancement of tissue-engineering has made possible dermal replacement on human wounds to facilitate healing.

A new sponge composed of collagen and glycosaminoglycans (chondroitins 4 and 6 sulphate), reticulated by ionic bonds with chitosan before freeze-drying, was developed in France. This sponge is a non-toxic product due to its non-chemical reticulation (ionic bonds), biocompatible and biodegradable processes, handling and storable easily.

The objective of this study is to demonstrate that such a substitute, cellularized by functional allogenic fibroblasts, and complying with all safety conditions, enables to lead to healing of diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patient aged ≥ 18
* Patient with documented and stable* type I or II diabetes mellitus
* With diagnosis of neuropathic foot ulcer located on the plantar surface of the forefoot
* Ulcer with a surface area comprised between 1 and 15 cm2 included (after mechanical debridement of the ulcer)
* Palpable pulse evidenced on both feet (presence of dorsalis pedis pulse and posterior tibial pulse) or in absence of one pulse, a Systolic Pressure Index (SPI) by Doppler > 0.9 on the target limb
* Presence of diabetic foot ulcer for at least 4 weeks prior to enrolment
* Patient's ulcer extending through the dermis without exposure of muscle, tendon, bone, or joint capsule *means confirmed by HbA1C at least every 4 months

Exclusion Criteria:

* Typical Charcot's foot
* Decrease or increase in the size of the ulcer by 50% or more during the run-in period
* Presence of osteitis (eq Br osteomyelitis) at the inclusion visit (evidenced with a radiological lesion facing the wound (bone erosion or disappearance of the cortical bone))
* Clinical evidence of Pedis grade 3, or 4 infection at the inclusion visit
* Patient who cannot have an off-loading method
* Patient with working activity who cannot be on sick-leave during the study period.
* Patient presenting a known allergy to collagen, streptomycin, penicillin and/or products of bovine origin
* Dialysed patient
* Patient suffering from a psychiatric disorder not treated
* Clinical evidence of gangrene on any part of the affected foot
* Patient receiving corticosteroids, NSAIDs, immunosuppressive or cytotoxic agents, all systemic agents that can affect wound repair or any treatment that might interfere with the assessment of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Complete wound closure at week 12 | 12 weeks

SECONDARY OUTCOMES:
Time to complete wound healing | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Chosidow, MD, PhD, Study Chair — Hôpital Tenon, Paris
Locations (7):
- France (7):
  - Marseille
  - Nancy
  - Nîmes
  - Paris
  - Roubaix
  - Thionville
  - Toulouse